CLINICAL TRIAL: NCT02028338
Title: Phase 2a Safety Study of a Vaginal Ring Containing Dapivirine in Adolescent Females
Brief Title: Study of Dapivirine Vaginal Ring (VR) in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Microbicide Trials Network (Network); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTN-023/IPM 030; 11927 (Other: DAIDS); DAID US NIAID (Other Grant/Funding Number: 3UM1AI068633-07S1 UM1 AI068615)
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapivirine ring (Experimental): dapivirine vaginal ring (25 mg)
  Interventions: Combination Product: dapivirine ring
- Placebo ring (Placebo Comparator): silicone vaginal ring
  Interventions: Combination Product: placebo ring

INTERVENTIONS:
Combination Product: placebo ring — intravaginal ring silicone elastomer intravaginal ring containing no drug product
  Arms: Placebo ring
Combination Product: dapivirine ring — intravaginal ring silicone elastomer intravaginal ring containing 25 mg dapivirine
  Arms: Dapivirine ring

SUMMARY:
To assess the safety of dapivirine (25 mg) administered via a silicone vaginal ring in HIV-uninfected adolescent females, when inserted once every 4 weeks during 24-week of study product use.

DETAILED DESCRIPTION:
MTN-023/IPM 030 is a Phase 2a, two-arm, placebo-controlled, double-blinded, multi-site, randomized trial of dapivirine vaginal ring (VR) versus placebo VR. The clinical trial is designed to assess the safety of dapivirine (25 mg) administered via a silicone vaginal ring (primary objective) and evaluate the acceptability of the dapivirine or placebo VR in sexually experienced, HIV-uninfected adolescent females, when inserted once every 4 weeks during 24-weeks of study product use.

Approximately 96 participants will be randomized in a 3:1 ratio to receive either a silicone elastomer vaginal ring containing 25 mg of dapivirine or a placebo VR. The ring will be replaced every 4 weeks during the 24 week study product use period.

Use of a VR to provide sustained delivery of microbicides is a novel investigational method for prevention of heterosexual transmission of HIV in women. This drug delivery method may circumvent potential difficulties related to adherence to daily or coitally-dependent uses of microbicide regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 through 17 years (inclusive) at Enrollment, verified per site SOPs
2. Able and willing to provide written informed assent/consent and able to obtain written parental or guardian permission (as specified in site SOP) to be screened for and to enroll in MTN-023/IPM 030
3. Able and willing to provide adequate locator information, as defined in site SOPs
4. Able to communicate in spoken and written English
5. Able and willing to comply with all study procedural requirements
6. Per participant report at Screening and Enrollment, willing to abstain from inserting anything into the vagina for 72 hours prior to each follow-up visit, including abstaining from penile-vaginal intercourse. Note: In the event the vaginal ring has been expelled and requires reinsertion, repositioning the vaginal ring is permitted
7. In general good health as determined by the Investigator of Record (IoR)/designee at Screening and Enrollment
8. Assessment of onset and progression of puberty, as measured by Tanner stage 4 or 5 at Screening, per participant report and/or clinician assessment
9. HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithm in Appendix II)
10. Per participant report at Screening, history of sexual intercourse (at least one episode in participant's lifetime)
11. Per participant report at Screening and Enrollment, agrees to use condoms for sexual intercourse
12. Negative pregnancy test at Screening and Enrollment
13. Per participant report, using an effective method of contraception for at least 30 days (inclusive) prior to Enrollment, and intending to continue use of an effective method for the duration of study participation; effective methods include:

    * hormonal methods (except contraceptive ring)
    * intrauterine device (IUD)
    * sterilization (of participant, as defined in site SOPs)
14. At Screening and Enrollment, participant states a willingness to refrain from inserting the following vaginal products and/or objects into the vagina; spermicides, diaphragms, contraceptive vaginal rings, menstrual cups, cervical caps (or any other vaginal barrier method), douches, lubricants, for the 5 days prior to Enrollment throughout the duration of study participation. Note: Neither the use of tampons or sex toys, nor participant engagement in coitus is restricted.
15. At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation, unless approved by the PSRT

Exclusion Criteria:

1. Per participant report at Screening, intends to do any of the following during the study participation period:

   1. become pregnant
   2. relocate away from the study site
   3. travel away from the study site for more than 4 consecutive weeks
2. Diagnosed with a urinary tract infection (UTI) and/or reproductive tract infection (RTI) at Screening and/or Enrollment. Note: Otherwise eligible participants diagnosed with UTI during Screening will be offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 56 days of obtaining informed consent for Screening, the participant may be enrolled.
3. Diagnosed with pelvic inflammatory disease and/or an sexually transmitted infection (STI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines within 60 days of Enrollment (inclusive)
4. At Enrollment, has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff)** Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary. Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved. If improvement to a non-exclusionary grade or resolution is documented within 56 days of providing informed consent for screening, the participant may be enrolled.
5. Participant report and/or clinical evidence of any of the following:

   1. Known adverse reaction to any of the study products (ever)
   2. Known HIV-infected partner
   3. Non-therapeutic injection drug use in the 12 months prior to Screening
   4. The use of HIV Post-exposure prophylaxis (PEP) and/or Pre-exposure prophylaxis (PrEP) within the 6 months prior to Enrollment
   5. Currently breastfeeding
   6. Last pregnancy outcome within 90 days or less of Screening
   7. Participation in any other research study involving drugs, medical devices, vaginal products, or vaccines, within 60 days of Screening
   8. Participant report of 3 or more penile-vaginal sexual partners in the month prior to Screening
   9. At Enrollment, as determined by the IoR/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
6. Has any of the following Grade 1 or higher* laboratory abnormalities at Screening Visit:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT)
   2. Creatinine
   3. Hemoglobin
   4. Platelet count Note: Otherwise eligible participants with an exclusionary test may be re-tested during the screening process. Please see the MTN-023/IPM 030 SSP for additional details.
7. Has any other condition that, in the opinion of the IoR/designee, would preclude informed assent/consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

   * Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009) **Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009)

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Alabama CRS 84519th street south, BBRB 203A, Birmingham, Alabama
  - The university of Colorado, 13123 E. 16th Ave., Box 025, Aurora, Colorado
  - The University of Colorado; 13123 E. 16th Ave., Box 025, Aurora, Colorado
  - The Fenway Institute, 1340 Boylston Street, Boston, Massachusetts
  - The Fenway Institute; 1340 Boylston Street, Boston, Massachusetts
  - Montefiore Medical Center, 3514 Wayne Ave, The Bronx, New York
  - Montefiore Medical Center; 3514 Wayne Ave, The Bronx, New York
  - University of Pittsburgh CRS, 3601 fifth Ave, Room 737, Pittsburgh, Pennsylvania
  - University of Pittsburgh CRS, 3601 Fifth Avenue, Room 737; Falk Medical Building,, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital 262 Danny Thomas PL., Memphis, Tennessee
  - St. Jude Children's Research Hospital; 262 Danny Thomas Pl., Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bunge KE, Levy L, Szydlo DW, Zhang J, Gaur AH, Reirden D, Mayer KH, Futterman D, Hoesley C, Hillier SL, Marzinke MA, Hendrix CW, Gorbach PM, Wilson CM, Soto-Torres L, Kapogiannis B, Nel A, Squires KE; MTN-023/IPM 030 Study Team. Brief Report: Phase IIa Safety Study of a Vaginal Ring Containing Dapivirine in Adolescent Young Women. J Acquir Immune Defic Syndr. 2020 Feb 1;83(2):135-139. doi: 10.1097/QAI.0000000000002244. PMID 31929401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As part of participant outreach and recruitment strategies, trial staff pre-screened potential trial participants at either on-site or off-site locations. During these interactions, trial staff explained the trial to potential participants, ascertained elements of presumptive eligibility.
Pre-assignment Details: Screening Visit were done up to 56 days prior to Enrollment Visit. Some cases, multiple visits were conducted to complete all screening procedures. Written informed participant assent and parental/guardian consent for screening were obtained.
  Participants who expressed an interest in involving her current sexual partner regarding trial participation was encouraged to bring her partner to the research center where a staff member explained the trial.
Period: Overall Study
Arm/Group | Dapivirine Ring | Placebo Ring
Started | 73 | 23
Completed | 69 | 22
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Unable to contact participant | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized 3:1
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapivirine Ring | Placebo Ring | Total
Number analyzed (Participants) | 73 | 23 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.3 (0.8) | 16.2 (0.7) | 16.3 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 23 | 96
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 4 | 20
  Not Hispanic or Latino | 57 | 19 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 13 | 47
  White | 20 | 4 | 24
  More than one race | 8 | 3 | 11
  Unknown or Not Reported | 10 | 1 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 23 | 96

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Dapivirine (25 mg) Administered Via a Silicone Vaginal Ring in HIV-uninfected Adolescent Females, When Inserted Once Every 4 Weeks During 24 Weeks of Study Product Use
Description: Grade 2 AEs as defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December 2004 (Clarification dated August 2009), Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies) judged to be related to IP.
  Grade 3 or higher AEs as defined by the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December 2004 (Clarification dated August 2009).
Time Frame: 6 months
Population: All participants randomized into the clinical trial were included in the primary analysis according to the principle of intent-to-treat (ITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Ring | Placebo Ring
Number analyzed (Participants) | 73 | 23
Participants
  Grade 2 Adverse Events related to IP | 8 | 2
  Grade 3 or higher events | 3 | 0

2. Secondary Outcome: The Acceptability of the Study VR (Dapivirine or Placebo) in HIV Uninfected Adolescent Females, When Inserted Once Every 4 Weeks for a 24 Week Period
Description: Participant's self-report on multiple components of acceptability via attitudinal questions (discreetness, likes and dislikes concerning the ring, attitude toward product characteristics, comfort and ease of use, partner reactions, and effect on sex) in categorical scales
Time Frame: 6 months
Population: The ITT population included all participants who were randomized to one of the two treatment groups, Dapivirine Vaginal Ring-004 or placebo ring. All participants who were included in a treatment group were analyzed as members of the group in which they were enrolled, regardless of adherence to the planned course of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Ring | Placebo Ring
Number analyzed (Participants) | 70 | 22
Participants
  Discreetness: number analyzed (Participants) | 48 | 13
  Discreetness: At least one negative report | 39 | 12
  Discreetness: All responses positive | 9 | 1
  Likes and dislikes concerning the ring: number analyzed (Participants) | 55 | 19
  Likes and dislikes concerning the ring: At least one negative report | 18 | 7
  Likes and dislikes concerning the ring: All responses positive | 37 | 12
  Attitude toward product characteristics: number analyzed (Participants) | 48 | 15
  Attitude toward product characteristics: At least one negative report | 14 | 4
  Attitude toward product characteristics: All responses positive | 34 | 11
  Comfort and ease of use: number analyzed (Participants) | 63 | 22
  Comfort and ease of use: At least one negative report | 27 | 10
  Comfort and ease of use: All responses positive | 36 | 12
  Partner reaction: number analyzed (Participants) | 28 | 8
  Partner reaction: At least one negative report | 12 | 3
  Partner reaction: All responses positive | 16 | 5
  Effect on sex: number analyzed (Participants) | 43 | 13
  Effect on sex: At least one negative report | 9 | 6
  Effect on sex: All responses positive | 34 | 7

3. Secondary Outcome: Adherence to the Study VR (Dapivirine or Placebo) in HIV Uninfected Adolescent Females, When Inserted Once Every 4 Weeks for a 24 Week Period
Description: Frequency of ring removals and expulsions based on the participant's self-report of ring use at monthly clinic visits according to the Ring Adherence CRF.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Ring | Placebo Ring
Number analyzed (Participants) | 73 | 23
Participants | 29 | 11

4. Secondary Outcome: The Systemic Dapivirine Exposure
Description: Dapivirine plasma concentrations measured at weeks 2, 4, 12 and 24.
Time Frame: 6 months
Population: The PK analysis population included all participants who were randomized to the Dapivirine Vaginal Ring-004 treatment group and had detectable dapivirine plasma or vaginal fluid concentrations at any time during follow-up.
Measure: Mean (Standard Deviation); unit: picograms/millilitre
Arm/Group | Dapivirine Ring
Number analyzed (Participants) | 73
picograms/millilitre
  Week 2 | 310.5 (102.0)
  Week 4 | 255.5 (91.1)
  Week 12 | 250.9 (96.6)
  Week 24 | 243.1 (116.3)

5. Secondary Outcome: Local Dapivirine Exposure
Description: Vaginal fluid dapivirine concentrations.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nanogram/milligram
Arm/Group | Dapivirine Ring
Number analyzed (Participants) | 73
nanogram/milligram
  Week 2 | 27.8 (22.7)
  Week 4 | 45.0 (40.9)
  Week 12 | 49.2 (53.6)
  Week 24 | 51.9 (58.2)

ADVERSE EVENTS:
Time Frame: 25 weeks
Description: Prior and concomitant medications were recorded at the Screening Visit and reviewed/updated at subsequent visits, and adverse events (AEs) were recorded after enrollment and recorded/updated at subsequent visits. Used rings were collected at the 4 Week, 8 Week, 12 Week, 16 Week, 20 Week, and 24 Week Visits.
Arm/Group | Dapivirine Ring | Placebo Ring
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/23
Other Adverse Events (participants affected / at risk) | 63/73 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapivirine Ring (N=73) | Placebo Ring (N=23)
Pelvic Inflammatory Disease (Renal and urinary disorders) | 1 | 0
Abdominal Incarcerated Hernia (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Ring (N=73) | Placebo Ring (N=23)
Ear Pain (Ear and labyrinth disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Bacterial vaginosis (Infections and infestations) | 9 | 2
Cystitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 4 | 0
Genitourinary chlamydia infection (Infections and infestations) | 8 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Pelvic Inflammatory disease (Infections and infestations) | 2 | 0 (0)
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 9 | 3
Viral infection (Infections and infestations) | 3 | 0
Viral Upper respiratory tract infection (Infections and infestations) | 3 | 0
Vulvovaginal candidiasis (Infections and infestations) | 7 | 3
Vulvovaginal Trichomonal (Infections and infestations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 1
Product Issue (Product Issues) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1
Breast tenderness (Reproductive system and breast disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 2
Menorrhagia (Reproductive system and breast disorders) | 5 | 2
Metrorrhagia (Reproductive system and breast disorders) | 15 | 6
Pelvic Pain (Reproductive system and breast disorders) | 7 | 0
Uterine spasm (Reproductive system and breast disorders) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 11 | 8
Vaginal Odour (Reproductive system and breast disorders) | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other